CLINICAL TRIAL: NCT01076374
Title: Medtronic Adapta/Versa/Sensia Long Term Reliability Study
Brief Title: MEDTRONIC ADAPTA, VERSA AND SENSIA nEw3 POST APPROVAL STUDY
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: nEw3 PAS
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Arrhythmia; Bradycardia
Keywords: pacemaker
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of this study is to assess the long term reliability of the Medtronic Adapta®/Sensia™/Versa™ platform of devices. This study is required by FDA as a condition of approval of nEw3 devices. Patients will be followed for 5 years after implant. This study utilizes data collected from the System Longevity Study (SLS).

DETAILED DESCRIPTION:
The rate of device malfunctions will be determined and a comparison to historical controls will be done.

ELIGIBILITY:
Inclusion Criteria:

* Subjects or appropriate legal guardians provide written informed consent and/or authorization for access to and use of health information, as required by an institution's IRB/MEC/REB.

AND one of the following must also apply:

* Subjects indicated for implant or within six months post-implant of a Medtronic market-released lead connected to a Medtronic Adapta®, Sensia™, or Versa™ IPG. The Medtronic lead must be used for pacing, sensing or defibrillation application.
* Subjects who participated in a qualifying study (IDE) of a Medtronic cardiac therapy product and: 1) have a Medtronic Adapta®, Sensia™, or Versa™ IPG 2)product is market-released 3) complete implant and follow-up data, including product-related adverse events are available and 4) subject of appropriate legal guardian authorizes release of subject study data to SLS
* Subjects implanted with a Medtronic Adapta®, Sensia™, or Versa™ IPG and Medtronic CapSure Epi Leads (model 4965 and 4968) at a minimum of three pre-selected sites to retrospectively collect data for post approval requirements.

Exclusion Criteria:

* Subjects who are, or will be inaccessible for follow-up at a SLS center
* Subjects with exclusion criteria required by local law (EMEA only)
* Subjects receiving an implant of a Medtronic device at a non-participating center and the implant data and current status cannot be confirmed within 30 days after implant
* Subjects implanted with a Medtronic device whose predetermined enrollment limit for that specific product has been exceeded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects implanted with a Medtronic Adapta®, Sensia™, or Versa™ IPG.
Sampling Method: Non-Probability Sample
Enrollment: 2927 (Actual)
Dates: Start 2008-07; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Rate of device malfunctions | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: nEw3 PAS Clinical Trial Leader, Study Chair — Medtronic
Locations (129):
- United States (110):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Gilbert, Arizona
  - Scottsdale, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Bakersfield, California
  - Chula Vista, California
  - Downey, California
  - East Palo Alto, California
  - La Jolla, California
  - Long Beach, California
  - Los Angeles, California
  - Redding, California
  - Salinas, California
  - San Diego, California
  - Santa Rosa, California
  - Torrance, California
  - Van Nuys, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Clearwater, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Tampa, Florida
  - Albany, Georgia
  - Atlanta, Georgia
  - Columbus, Georgia
  - Marietta, Georgia
  - Oak Lawn, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Edgewood, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Alexandria, Louisiana
  - Baton Rouge, Louisiana
  - Covington, Louisiana
  - Salisbury, Maryland
  - Silver Spring, Maryland
  - Takoma Park, Maryland
  - Towson, Maryland
  - Worcester, Massachusetts
  - Lansing, Michigan
  - Marquette, Michigan
  - Saginaw, Michigan
  - Ypsilanti, Michigan
  - Coon Rapids, Minnesota
  - Minneapolis, Minnesota
  - Robbinsdale, Minnesota
  - Rochester, Minnesota
  - Saint Louis Park, Minnesota
  - Saint Paul, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - Washington, Missouri
  - Lebanon, New Hampshire
  - Browns Mills, New Jersey
  - Ocean City, New Jersey
  - Parlin, New Jersey
  - West Orange, New Jersey
  - Albuquerque, New Mexico
  - Garden City, New York
  - Henderson, New York
  - Huntington, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - Utica, New York
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Sayre, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Florence, South Carolina
  - Sioux Falls, South Dakota
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Burlington, Vermont
  - Chesapeake, Virginia
  - Fairfax, Virginia
  - Olympia, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Linz, Austria
- Hasselt, Belgium
- Canada (6):
  - Calgary, Alberta
  - Kingston, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Regina, Saskatchewan
- Copenhagen, Denmark
- France (2):
  - Marseille
  - Nantes
- Homburg/Saar, Germany
- Italy (2):
  - Reggio Emilia
  - Udine
- Netherlands (2):
  - Eindhoven
  - Rotterdam
- Belgrade, Serbia
- Skövde, Sweden
- Zurich, Switzerland